CLINICAL TRIAL: NCT02328274
Title: A Modified Technique for Laparoscopic Subtotal Hysterectomy
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Chen Chuang, M.D, Far Eastern Memorial Hospital
Other Study IDs: 103138-E
Record Dates: First submitted 2014-12-25; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Subtotal Hysterectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: A Modified Technique for Laparoscopic Subtotal Hysterectomy — incorporation of two methods of vessels ligation and laparoscopic in situ morcellation

SUMMARY:
Laparoscopic subtotal hysterectomy (LASH) for benign uterine lesion has regained its popularity in the past decade due to its minimal invasiveness that results in less operation time, less blood loss and quicker return to normal activity. The standard surgical procedure in LASH includes separation of adnexa and round ligament from pelvic sidewall or uterus, dissection of the vesico-uterine peritoneum and opening of the paravesical space; followed by amputation of the uterus with energy-producing modalities (such as Harmonic Scalpel, monopolar electrocautery, bipolar electrocautery). Large uteri may result in longer operative time and higher possibility of conversion to laparotomy due to technical difficulty and excessive blood loss. In order to overcome these difficulties, we introduce a modified surgical technique of LASH which incorporated two methods of vessels ligation and laparoscopic in situ morcellation.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 20 years old and above with symtomatic uterine myomas or adenomyosis
* complete medical record

Exclusion Criteria:

* patients aged below 20 years old
* uterine malignancy
* incomplete medical record

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients aged 20 years old and above with symtomatic uterine myomas or adenomyosis
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Operation time | at time of surgery
Intraoperative blood loss | at time of surgery

SECONDARY OUTCOMES:
Post-operative complications | up to 7 days post operation
  such as ureteral injury, bowel perforation, conversion to laparotomy, recurrent vaginal bleeding